CLINICAL TRIAL: NCT05706870
Title: A Multicenter Randomized Double-blind Placebo-controlled Parallel Group Phase II Study Evaluating the Clinical Efficacy and Safety of GN-037 Cream Used in the Treatment of Mild to Moderate Plaque Psoriasis
Brief Title: Phase II Study Evaluating the Clinical Efficacy and Safety of GN-037 in Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GEN İlaç ve Sağlık Ürünleri A.Ş. (Industry)
Collaborators: Monitor CRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MON886.151.7
Record Dates: First submitted 2023-01-10; First posted 2023-01-31 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis
Keywords: mild to moderate plaque psoriasis; local treatment
MeSH Terms: conditions — Psoriasis | interventions — Clobetasol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GN-037 cream (Experimental): Psoriatic patients will receive GN-037 cream in 2:2:1 ratio
  Psoriatic patients will receive GN-037 cream twice daily on a selected body target lesion
  GN-037 cream will be applied as a thin film layer for 4 weeks.
  Interventions: Drug: GN-037
- Clobetasol 17-propionate cream (Active Comparator): Clobetasol 17-propionate cream will be applied in 2:2:1 ratio
  Psoriatic patients will receive clobetasol 17-propionate cream twice daily on a selected body target lesion
  Clobetasol 17-propionate will be applied as a thin film layer for 4 weeks.
  Interventions: Drug: Clobetasol 17-propionate
- Placebo (Placebo Comparator): Placebo cream will be applied in 2:2:1 ratio
  Psoriatic patients will receive placebo cream twice daily on a selected body target lesion
  Placebo cream will be applied as a thin film layer for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GN-037 — GN-037
  Arms: GN-037 cream
Drug: Clobetasol 17-propionate — Clobetasol 17-propionate
  Arms: Clobetasol 17-propionate cream
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This Phase II study was designed as a multicenter, randomized, double-blind, placebo-controlled and 3-parallel arm, to assess clinical efficacy, safety, and tolerability of GN-037 versus clobetasol 17-propionate and placebo in patients diagnosed with mild to moderate plaque psoriasis at least 6 months ago

DETAILED DESCRIPTION:
A total of 190 patients aged between 18-65 years diagnosed with plaque psoriasis are planned to be included in the study. The study consists of three periods:

Screening period: Within 4 weeks before baseline visit (-28 days to 0 days)

Treatment period: 4 weeks

Follow-up period with observation: 4 weeks

The study is planned to last a maximum of 12 weeks for each patient. Study consists of 5 visits: baseline (day 1), week 2, week 4, week 6 and week 8 which is a follow-up period with observation.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 18-65
2. Patients who can give their written informed consent prior to initiating any evaluation or procedure related to the study.
3. Patients with negative SARS-CoV-2 PCR test result
4. Patients who were diagnosed with mild or moderate plaque psoriasis at least 6 months ago by a dermatologist and whose diagnosis was confirmed according to the clinical judgment of the research physician at the time of enrolment.
5. Patients with a Investigator Global Assessment (IGA) score of 2 or 3 at the screening visit [Face, scalp, palms, soles, armpits, and intertriginous areas will be excluded from this assessment]
6. Patients with plaque psoriasis lesions covering a body surface area (BSA) of at least 3% to 12% [Face, scalp, palms, soles, axillae, and intertriginous areas will be excluded from this assessment.]
7. Patients who received the last psoriasis treatment 4 weeks or before
8. Patients who are confirmed to be healthy by medical history and physical examination and who do not have any clinically significant disease/condition other than plaque psoriasis that, at the discretion of the investigator, could affect the study evaluation.
9. Patients who can protect the lesion areas from ultraviolet (UV) rays (natural or artificial) during the study
10. Female patients: Patients who had a negative pregnancy test at the screening visit, did not breastfeed, did not plan pregnancy during the study, and agreed to use an effective method of contraception until the end of the study.

    Male patients: Patients who agreed to use an effective method of contraception for the duration of the study.
11. Patients who can comply with all scheduled visits, laboratory tests, and other study procedures
12. Patients with normal adrenocorticotropic hormone (ACTH) stimulation test
13. Patients with normal dihydroepiandrostenedione sulfate (DHEAS) levels

Exclusion Criteria:

1. Patients with a known sensitivity/hypersensitivity to any component of the drugs to be used in the study
2. Pregnant or lactating or female patients with a positive pregnancy test
3. Patients who are resistant/unresponsive to corticosteroids
4. Patients with psoriasis (eg guttate, erythrodermic, exfoliative or pustular) that, in the opinion of the investigating physician, resolves spontaneously or rapidly worsens
5. Patients with other inflammatory skin disease (eg, atopic dermatitis, contact dermatitis, eczema, tinea corporis) that, in the opinion of the investigative physician, may affect study evaluations at the targeted treatment sites
6. Patients who received phototherapy, photochemotherapy, systemic or local treatment for psoriasis or used systemic anti-inflammatory agents in the last 4 weeks
7. Patients who received biologic therapy for psoriasis in the last 3 months
8. Immunosuppressive or immunocompromised patients (patients who have taken immunosuppressive drugs in the last 2 months will also be excluded)
9. Patients who have received any cancer treatment in the last 1 year
10. Patients with severe hypertension (systolic blood pressure [SBP] > 160 mmHg or diastolic blood pressure [DBP] > 100 mmHg)
11. Patients who cannot comply with the study procedures/rules and cannot be in harmony with the research team
12. Patients who have participated in another clinical trial in the last 2 months or who are taking part in another clinical trial concurrently
13. Patients with a known abnormality of the hypothalamus-pituitary-adrenal axis (HPA axis)
14. Patients using products containing dihydroepiandrostenedione (DHEA) or dihydroepiandrostenedione sulfate (DHEAS) in the last 1 month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Improvement in Investigator Global Assessment (IGA) score evaluated at weeks 2, 4, 6 and 8 in each arm. | 28 days
  Improvement will be evaluated as the number and percent of patients with at least 2 points improvement in IGA score, and IGA score equating to 0 or 1.

SECONDARY OUTCOMES:
Mean change in %BSA affected from baseline at weeks 2, 4, 6 and 8 in each arm. | 28 days
  Target plaque area (cm2) was determined by multiplying the longest diameter (cm) of the target plaque by the widest perpendicular diameter (cm). A negative percent change indicates a mild disease.
Improvement in Psoriasis Area Severity Index (PASI) from baseline at weeks 2, 4, 6 and 8 in each arm. Improvement will be evaluated as the number and percent of patients with ≥75% improvement in PASI score. | 28 days
  The PASI scoring system takes into account the overall severity of erythema (redness), induration (plaque thickness) and scaling, and the extent of %Body Surface Area affected with psoriasis. Higher scores indicate more severe disease. PASI is a static assessment made without reference to previous scores.
Mean change in in total plaque severity score (TPSS) from baseline at week 2, 4, 6 and 8 in each arm. | 28 days
  For TPSS, all target lesions were scored individually for signs of induration, scaling, and erythema using a 5-point severity scale: 0 = none; 1 = mild; 2 = moderate; 3 = severe; 4 = very severe. A negative percent change indicates better outcome.
Improvement in target lesion healing from baseline at weeks 2, 4, 6 and 8 in each arm. | .28 days
  Improvement will be evaluated as the number and percent of patients whose target lesion erythema, plaque thickness and scaling score improvement at least 2 points at week 2, 4, 6 and 8 compared to baseline in each arm. Additionally, at which week at least 50% improvement in the target lesion healing is observed in each arm will be evaluated.
  Target plaque area (cm2) was determined by multiplying the longest diameter (cm) of the target plaque by the widest perpendicular diameter (cm).
Improvement in Dermatology Life Quality Index (DLQI) | 28 days
  Improvement in DLQI at weeks 4 and 8 compared to baseline.
Safety, Adverse Events and Serious Adverse Events | 56 days
  Safety will be evaluated as the number and ratio of patients with adverse events and serious adverse events in each arm. Additionally, number of adverse events which resulted in discontinuation of the study treatment in each arm will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Nadir Ulu, MD PhD, Study Chair — Gen Ilac
Locations (18):
- Turkey (Türkiye) (18):
  - Ankara Etlik City Hospital, Ankara
  - Balıkesir University Faculty of Medicine, Balıkesir
  - Uludag University Faculty of Medicine, Bursa
  - Pamukkale University Faculty of Medicine, Denizli
  - Ataturk University Research Hospital, Erzurum
  - Istanbul University Cerrahpasa Faculty of Medicine, Istanbul
  - Basaksehir Cam and Sakura City Hospital, Istanbul
  - Bezmialem Vakif University Faculty of Medicine, Istanbul
  - Haydarpasa Numune Training and Research Hospital, Istanbul
  - Istanbul Haseki Training and Research Hospital, Istanbul
  - Istanbul University Istanbul Faculty of Medicine, Istanbul
  - University of Health Sciences Bakırkoy Dr. Sadi Konuk Training and Research Hospital, Istanbul
  - İzmir Democracy University Buca Seyfi Demirsoy Training And Research Hospital, Izmir
  - Erciyes University Faculty of Medicine, Kayseri
  - Necmettin Erbakan University Meram Faculty of Medicine, Konya
  - Mersin University Faculty of Medicine, Mersin
  - Samsun Ondokuz Mayis University Faculty of Medicine, Samsun
  - Uşak Training and Research Hospital, Uşak

REFERENCES:
- [Derived] Engin B, Guler Ozden M, Karstarli Bakay OS, Kartal SP, Zindanci I, Cinar SL, Dursun R, Pehlivan Ulutas G, Ozkok Akbulut TO, Hapa FA, Bulbul Baskan E, Melikoglu M, Polat Ekinci A, Demirel Ogut N, Hizli P, Turkoglu Z, Kucuk OS, Topkarci Z, Tursen U, Canpolat F, Ucgun H, Yasar S, Temiz SA, Dogramaci AC, Altug S, Kozlu S, Ulu N, Serdaroglu S. A Multicenter Randomized Double-Blind Vehicle-Controlled Parallel Group Phase 2 Study Evaluating the Efficacy and Safety of GN-037 Cream in Patients with Mild-to-Moderate Plaque Psoriasis. Dermatol Ther (Heidelb). 2024 Dec;14(12):3337-3350. doi: 10.1007/s13555-024-01301-1. Epub 2024 Nov 22. PMID 39578347
- [Derived] Sezer Z, Inal A, Cinar SL, Mazicioglu MM, Altug S, Karasulu HY, Diril M, Mehmetoglu Al A, Kozlu S, Ulu N. Safety and Efficacy of a Novel Combination Cream (GN-037) in Healthy Volunteers and Patients with Plaque Psoriasis: A Phase 1 Trial. Dermatol Ther (Heidelb). 2023 Jul;13(7):1489-1501. doi: 10.1007/s13555-023-00939-7. Epub 2023 Jun 10. PMID 37300792